CLINICAL TRIAL: NCT03459287
Title: A Randomized, Double-Blinded, Controlled, Parallel Group, Non-inferiority, Phase III Study to Evaluate the Efficacy and Safety of the INTERCEPT Blood System for Red Blood Cells in Patients Undergoing Complex Cardiac Surgery Procedures
Brief Title: Study to Evaluate the Efficacy & Safety of the INTERCEPT Blood System for RBCs in Complex Cardiac Surgery Patients
Acronym: ReCePI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cerus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLI 00125
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-06

CONDITIONS: Anemia
Keywords: INTERCEPT; Red Blood Cells; RBC; Pathogen Inactivation; Cerus; Pathogen Reduction; Cardiovascular surgery
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Intervention Model Description: Parallel group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- INTERCEPT (test) (Experimental): The INTERCEPT treatment process uses amustaline and glutathione together with a processing solution in a single-use disposable set and results in pathogen and leukocyte inactivated RBCs suspended in SAG-M additive solution (INTERCEPT RBCs). The INTERCEPT treatment will be performed on leukocyte reduced RBC components prepared from whole blood collections and suspended in AS-5 additive solution within 24 hours of collection. The test component is allogeneic INTERCEPT RBCs suspended in SAG-M and stored at 1°C to 6 for up to 35 days post-donation and administered intravenously. Dose and schedule of RBC transfusions will be determined by the treating physician.
  Interventions: Device: INTERCEPT
- Conventional (Control) (Active Comparator): The control transfusion component is a conventional leukocyte-reduced RBC component in an FDA approved additive solution (AS-1, AS-3 or AS-5) stored at 1°C to 6°C for up to 35 days post-donation and administered intravenously. The Control RBC components will be handled and labeled in a manner so as to maintain blinding. Dose and schedule of RBC transfusions will be determined by the treating physician.
  Interventions: Device: Control

INTERVENTIONS:
Device: INTERCEPT — Pathogen reduced RBCs
  Arms: INTERCEPT (test)
Device: Control — Conventional RBCs
  Arms: Conventional (Control)

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of RBC transfusion for support of acute anemia in cardiovascular surgery patients based on the clinical outcome of renal impairment following transfusion of red blood cells (RBCs) treated with the INTERCEPT Blood System (IBS) for Red Blood Cells compared to patients transfused with conventional RBCs.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, double-blinded, active controlled, parallel-design, non-inferiority study.

Screening/Recruitment

In order to minimize the number of patients who enroll in the study but do not require RBC transfusion, only patients with a relatively high likelihood to receive a RBC transfusion as determined by the Investigator (e.g., patients receiving aspirin, clopidogrel (or analogs) and/or GPIIb/IIIa inhibitors), or patients with a TRUST Score of ≥3 will be eligible for enrollment. Patients ≥11 years of age undergoing complex cardiac surgery may be identified through pre-operative scheduling procedures in advance of their surgery.

Patients undergoing urgent or emergent cardiac surgery are eligible for the study, subject to institutional review board (IRB) approval of an appropriate informed consent process.

All potentially eligible patients will be approached for study consent/assent within 30 days prior to their surgical procedure. Subjects who consent/assent to the study will be assigned a subject ID number and undergo screening.

Screening will include documentation of the patient's pre-surgical exposure to radiographic contrast media and number of prior pregnancies (females). Screening data may be derived from the medical record when performed within 30 days prior to their surgical procedure. Eligibility status and other study data including all TRUST components will be entered into the clinical database via an electronic data capture (EDC) system using electronic case report forms (eCRFs). Patients who fail eligibility for any or multiple inclusion/exclusion criteria may be rescreened for eligibility closer to the time of surgery.

Randomization and Blinding

Eligible subjects will be randomized up to 7 days before or on the day of scheduled surgery (Day 0). An Interactive Web Response System (IWRS) will be used for electronic randomization of eligible patients. Randomization (in 1:1 ratio for Test:Control) stratified by site, pre-existing renal impairment (baseline sCr ≥1.2 mg/dL vs. < 1.2 mg/dL), and cardiac surgery group (more at risk for renal complications vs. less at risk) will be employed. Screened subjects who receive a red cell transfusion prior to randomization will no longer be considered for randomization, and their participation in the study will end. Patients may be rescreened for eligibility closer to the time of surgery.

Treatment

Once a subject is randomized, only study RBCs (Test or Control, per the subject's randomization) should be dispensed and transfused during the acute transfusion support period (Day 0 to Day 7 post surgery, hospital discharge, or death, whichever is first), as clinically indicated and determined by the treating physician.

In rare exceptions where study RBCs are unavailable or patient's need for RBC transfusions exceeds the quantity of study RBCs in inventory at the hospital blood bank (e.g., during a Massive Transfusion Protocol), a transfusion using non-study RBC (conventional) may be given to provide the patient with an appropriate and necessary treatment. In this case, a protocol deviation should be documented. If a study RBC transfusion is given after randomization before surgery commences, a protocol deviation should also be documented.

Treatment assessments will be divided into an acute transfusion support period starting the day of surgery (Day 0 up to Day 7) during which study RBC (Test or Control) are administered, a post-surgical follow-up period of a minimum of 28 days after the last study transfusion to collect additional safety data, a clinical assessment at day 30 after surgery specifically for mortality and RRT status, and a visit at day 75 (±15) after the last study transfusion to assess mortality and RRT status, and collect samples for serological screening for antibodies specific to INTERCEPT RBCs.

In all patients, anesthesia and surgical procedures will be performed according to the local standards of care. Following the acute transfusion support period, subjects may receive conventional RBC components if additional transfusions are needed, as indicated by their treating physician.

Study Assessments: Monitoring and Follow-up

Baseline through Acute Transfusion Support Period (Pre-Op Day -1 up to Post-Op Day 7):

A screen for antibodies specific for INTERCEPT RBCs should be performed every time that a routine IAT is performed during the acute 7-day study transfusion period.

A blood sample for sCr will be taken at 48 ±4 hours after completion of surgery for both transfused and non-transfused subjects., A sCr will be determined on a daily basis during the acute transfusion support period up to 7 days post-surgery. Other parameters including additional sCr will be collected on eCRFs only when available in the medical record.

Randomized subjects who do not receive an RBC transfusion following randomization within the first 48 hours after surgery will be discontinued from the study and replaced.

Daily sCr assessments will be recorded up to and including 48 ±4 hours for transfused and non-transfused subjects. Other post baseline laboratory parameters and adverse events (AEs) will not be collected for non-transfused subjects. Vital status will be reported for randomized and non-transfused subjects at the time of discontinuation.

Hemodynamic and laboratory measures will be assessed pre-operatively (Day -1, Baseline) and daily as available in the medical record from post operative Day 1 through Day 7, hospital discharge or death, whichever occurs first. If a subject is discharged prior to Day 7 but returns to the study site for a standard of care visit on Day 7, blood samples should be obtained on that day for a complete blood count and sCr determination.

Hemodynamic parameters that will be collected if available, include heart rate, blood pressure, mean arterial pressure, central venous pressure (CVP), and peripheral oxygen saturation via pulse oximetry probe.

Laboratory parameters that will be captured on eCRFs include BUN, creatinine (sCr), AST, ALT, fibrinogen, bilirubin, troponin, hemoglobin, and platelet counts.

Transfusion reactions (TRs), adverse events (AEs) and serious adverse events (SAEs) will be assessed on a daily basis and documented in the eCRF from the start of surgery or the start of the first study transfusion (whichever is first) through post-operative Day 7 and as available through day 28 after the last study transfusion. Vital status will be reported for randomized and non-transfused subjects at the time of discontinuation.

NOTE: The following applies to randomized transfused subjects only.

Post-operative Day 8 (or Post-discharge, if earlier) through 28 Days After Last Study Transfusion:

Subjects will be monitored for TRs, AEs and SAEs following the 7-day acute transfusion support period, through 28 days after the last study transfusion or death, whichever occurs first, according to the local standard of care. In an outpatient setting, weekly telephone surveillance calls to the subject will be performed in order to collect safety events until the next follow-up visit.

28 (±3) Days After Last Study Transfusion or Premature Discontinuation from study:

Subjects who have been discharged should be scheduled for the follow up visit 28 (±3) days after the last study transfusion to obtain additional safety information, including patient-reported AEs/ SAEs; laboratory results including sCr, DAT/ IAT; a sample for HLA antibodies and antibodies specific to INTERCEPT RBCs will be obtained. All randomized subjects who receive any study RBC transfusion must have their vital status documented at this visit, or earlier, if the subject dies prior to the visit. If a subject has been discharged, other safety information (e.g., AEs and SAEs) may be obtained through medical records, the subject's physician, or a telephone interview with either the subject or a family member.

30 Days After Surgery:

All randomized subjects who receive a study RBC transfusion must have their vital status and need for RRT (defined as hemodialysis or peritoneal dialysis) documented at Day 30 after surgery. RRT that is provided prophylactically during surgery while patient is on a bypass machine (the pump), does not meet this endpoint. The vital status and RRT assessment on Day 30 can be performed either from the medical records, from a phone call to the subject or family, or during the visit 28±3 days after the last study transfusion (only if the last study transfusion was given at day 2 or later in the acute transfusion support period).

End of Study: 75 (±15 Days) After last Study Transfusion:

75 (±15) days after the last study transfusion (End of Study), serum samples for antibodies specific for INTERCEPT RBCs will be obtained, either in hospital, at a clinic visitor or offsite. Mortality and the need for RRT will be assessed

Data and Safety Monitoring Board (DSMB)

The study data and safety will be monitored by an independent Data and Safety Monitoring Board (DSMB). The primary mission of the DSMB is to ensure patient safety and protocol compliance for data collection. The DSMB will be assembled by the Sponsor and composed of transfusion medicine and other experts as per the DSMB charter. DSMB members will be independent of the Sponsor.

Interim Analysis and Early Stopping Rule

Aside from the blinded interim analysis for sample size re-estimation performed in October 2021, no other interim analysis is planned for this study to compare treatment differences with respect to efficacy or safety at any time prior to the completion of the study. Specific stopping rules, defined for safety considerations, are defined in Section 4.6 of the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 11 years of age
2. Weight ≥ 40 kg
3. Scheduled complex cardiac surgery or thoracic aorta surgery. The procedure may be performed either on or off cardiopulmonary bypass machine (CBP or "pump"). For the purposes of this protocol "Repeat procedure" means that the subject had a previous cardiac surgery. Procedures that qualify as complex cardiac surgery include but are not limited to, the following:

   * Single Vessel Coronary Artery Bypass Graft, first or repeat procedure
   * Multiple Coronary Artery Bypass Grafts, first or repeat procedure
   * Single Valve Repair or Replacement, first or repeat procedure
   * Multiple Valve Repair or Replacement, first or repeat procedure
   * Surgery involving both Coronary Artery Bypass Graft(s) and Valve Repair(s), first or repeat procedure
   * One or more of the following procedures, with or without Coronary Bypass Graft(s):

     * left ventricular aneurysm repair
     * ventricular and/or atrial septal defect repairs
     * Batista procedure (surgical ventricular remodeling)
     * surgical ventricular restoration
     * congenital cardiac defect repair
     * aortic procedures
     * other cardiac surgery or thoracic aorta surgery types with a high probability of bleeding
4. TRUST probability score (Alghamdi, Davis et al. 2006) ≥ 3, or currently on a regimen of aspirin (any dose), clopidogrel (or analogs) and/or GPIIb/IIIa inhibitors or at a high probability for need of a transfusion during or after surgery at the discretion of the Investigator
5. Female subjects of child-bearing potential must meet the 2 criteria below at screening:

   * Negative serum or urine pregnancy test
   * Use at least one method of birth control that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomized partner
6. Signed and dated informed consent/assent form

Exclusion Criteria:

1. Confirmed positive baseline serum/plasma antibody specific to INTERCEPT RBCs (S-303 specific antibody) screening panel prior to randomization.
2. Pregnant or breast feeding
3. Refusal of blood products or other inability to comply with the protocol in the opinion of the Investigator or the treating physician
4. Treatment with any medication that is known to adversely affect RBC viability, such as, but not limited to dapsone, levodopa, methyldopa, nitrofurantoin, and its derivatives, phenazopyridine and quinidine.
5. Planned cardiac transplantation
6. Active autoimmune hemolytic anemia
7. Left ventricular assist device (LVAD) or extracorporeal membrane oxygenation (ECMO) support pre operatively or planned need post-operatively
8. Cardiogenic shock requiring pre-operative placement of an intra-aortic balloon pump (IABP) (NOTE: IABP done for unstable angina or prophylactically for low ejection fraction is not excluded).
9. Planned use of autologous or directed donations.
10. RBC transfusion during current hospitalization prior to enrollment and randomization (within 7 days).
11. Participation in an interventional clinical study concurrently or within the previous 28 days. This includes investigational blood products, pharmacologic agents, imaging materials (including dyes), surgical techniques, or devices. Observational studies of FDA cleared or approved products or nutrition, psychology, or socioeconomic issues are not grounds for exclusion
12. Patients with a current diagnosis of either chronic kidney disease or acute kidney injury and with sCr ≥1.8 mg/dL at screening and patients requiring RRT. (NOTE: If sCr at screening is <1.8 mg/dL, a patient with a diagnosis of chronic or acute kidney injury alone is not excluded).
13. Patients with a current diagnosis of either chronic or acute hepatic insufficiency and with a total serum bilirubin ≥ 2.0 mg/dL (≥34.2 µmol/L). (NOTE: If total serum bilirubin at screening is <2.0 mg/dL, a patient with a diagnosis of chronic or acute hepatic failure alone is not excluded).
14. Pre-existing antibody(ies) to RBC antigens that may make the provision of compatible study RBC components difficult.
15. History of TRs requiring washed RBCs, volume reduced RBC, or RBCs with additive solution removed.
16. Patients with documented IgA deficiency or a history of severe allergic reactions to blood products.
17. Patients who require gamma-irradiated RBC blood components.
18. Positive DAT as defined below:

A polyspecific DAT reaction strength > 2+, or

A polyspecific DAT (any strength) in conjunction with pan-reactivity with a commercial IAT antibody screening panel that precludes the identification of underlying alloantibodies or indicates the presence of autoantibody

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2024-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Benjamin, MD, Principal Investigator — Cerus Corporation
Locations (18):
- United States (18):
  - University of California Los Angeles, Los Angeles, California
  - Stanford, Stanford, California
  - University of Colorado Hospital, Aurora, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Emory, Atlanta, Georgia
  - University of Kentucky, Lexington, Kentucky
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Mayo-Rochester, Rochester, Minnesota
  - Duke University Health System, Durham, North Carolina
  - Temple, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Texas Southwestern, Dallas, Texas
  - Houston Methodist, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Submit protocol, SAP and ICF.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Sekela ME, Snyder EL, Welsby IJ, Toyoda Y, Alsammak M, Sodha NR, Beaver TM, Pelletier JPR, Gorham JD, McNeil JS, Sniecinski RM, Pearl RG, Nuttall GA, Sarode R, Reece TB, Benjamin RJ; and the ReCePI Study Collaborators. Transfusion of Amustaline/Glutathione Pathogen-reduced Red Blood Cells in Cardiac Surgery: A Randomized Phase 3 Clinical Trial. Anesthesiology. 2025 Nov 1;143(5):1196-1210. doi: 10.1097/ALN.0000000000005716. Epub 2025 Aug 12. PMID 41085306
- [Derived] Karim C, Panigrahi A, Pearl RG, Sodha NR, Beaver TM, Pelletier JPR, Nuttall GA, Reece TB, Erickson A, Hedrick T, Liu K, Bentow S, Corash L, Mufti N, Varrone J, Benjamin RJ. Characterizing the antibody response to amustaline/glutathione pathogen-reduced red blood cells. Transfusion. 2025 Feb;65(2):344-353. doi: 10.1111/trf.18117. Epub 2024 Dec 25. PMID 39719927

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 636 subjects consented, 16 subjects did not meet inclusion criteria; 28 subjects met exclusion criteria; 11 other (surgery cancelled, subject chose not to be randomized), 581 subjects enrolled.
Period: Overall Study
Arm/Group | INTERCEPT (Test) | Conventional (Control)
Started | 296 | 285
Completed | 136 | 136
Not Completed | 160 | 149

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | INTERCEPT (Test) | Conventional (Control) | Total
Number analyzed (Participants) | 296 | 285 | 581
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 128 | 136 | 264
  >=65 years | 168 | 149 | 317
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.4 (13.1) | 63.2 (12.7) | 63.8 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 112 | 234
  Male | 174 | 173 | 347
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 14 | 27
  Not Hispanic or Latino | 282 | 271 | 553
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 31 | 28 | 59
  White | 258 | 245 | 503
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 4 | 6 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 296 | 285 | 581

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Have Received at Least One Study Transfusion With a Diagnosis of Renal Impairment Defined as:
Description: Any raised serum creatinine (sCr) level, occurring after transfusion of a study RBC, of ≥0.3 mg/dL (or 26.5 µmol/L) from the pre-surgery baseline within 48±4 hours of the end of surgery.
Time Frame: Within 48±4 hours of the end of surgery
Population: Participants who received at least one study transfusion with available data on the outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | INTERCEPT (Test) | Conventional (Control)
Number analyzed (Participants) | 157 | 161
Participants | 46 | 45

2. Primary Outcome: Percentage of Patients With Related Adverse Events
Description: Percentage of patients with any treatment-emergent adverse events (TEAEs) possibly, probably or definitely related to study RBC transfusion through 28 days after the last study transfusion.
Time Frame: From the start of the first study transfusion to 28 days after the last study transfusion (between 29 and 35 days depending on the day of the last study transfusion).
Population: Participants who received at least one study transfusion with available data on the outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | INTERCEPT (Test) | Conventional (Control)
Number analyzed (Participants) | 159 | 162
Participants | 4 | 1

3. Primary Outcome: Percentage of Patients With Treatment Emergent Antibodies
Description: Percentage of patients with treatment-emergent antibodies with confirmed specificity to INTERCEPT RBCs by the end of study.
Time Frame: From the start of the first study transfusion to 75 days after the last study transfusion (between 76-82 days depending on the day of the last study transfusion).
Population: Participants who received at least one study transfusion with available data on the outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | INTERCEPT (Test) | Conventional (Control)
Number analyzed (Participants) | 159 | 162
Participants | 5 | 0

4. Secondary Outcome: Percentage of Patients With a Diagnosis of Stage I, II or III Acute Kidney Injury
Description: The percentage of patients with a diagnosis of stage I, II, or III Acute Kidney Injury (KDIGO 2012) by day 7 post surgery, as defined by the change in serum creatinine (sCr) from baseline and the need for renal replacement therapy, i.e. clinical worsening of outcome from Stage I to Stage III. Stage I: sCr 1.5-1.9 times baseline within 7 days after surgery or > or=0.3 mg/dl (> or= 26.5 micromol/L) increase within 48 hrs of surgery; Stage II: sCr 2.0-2.9 times baseline within 7 days after surgery; Stage III: sCr 3.0 times baseline within 7 days after surgery or increase in sCr to > or=4.0 mg/dl (> or=353.6 micromol/L) or initiation of renal replacement therapy.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Groups:
- Test: The INTERCEPT treatment process uses amustaline and glutathione together with a processing solution in a single-use disposable set and results in pathogen and leukocyte inactivated RBCs suspended in SAG-M additive solution (INTERCEPT RBCs). The INTERCEPT treatment will be performed on leukocyte reduced RBC components prepared from whole blood collections and suspended in AS-5 additive solution within 24 hours of collection. The test component is allogeneic INTERCEPT RBCs suspended in SAG-M and stored at 1°C to 6 for up to 35 days post-donation and administered intravenously. Dose and schedule of RBC transfusions will be determined by the treating physician.
  INTERCEPT: Pathogen reduced RBCs
- Control: The control transfusion component is a conventional leukocyte-reduced RBC component in an FDA approved additive solution (AS-1, AS-3 or AS-5) stored at 1°C to 6°C for up to 35 days post-donation and administered intravenously. The Control RBC components will be handled and labeled in a manner so as to maintain blinding. Dose and schedule of RBC transfusions will be determined by the treating physician.
  Control: Conventional RBCs
Arm/Group | Test | Control
Number analyzed (Participants) | 159 | 162
Participants
  Diagnosis of KDIGO Stage II | 8 | 9
  Diagnosis of KDIGO Stage III | 15 | 7
  Diagnosis of KDIGO Stage I | 36 | 39

5. Secondary Outcome: Mortality or the Need for RRT
Description: Mortality or the need for RRT by 30 days post surgery
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | INTERCEPT (Test) | Conventional (Control)
Number analyzed (Participants) | 159 | 162
Participants | 16 | 8

6. Other Pre Specified Outcome: Number of Participants With Treatment-emergent (TE) Immunization to RBC Alloantigens
Description: Treatment-emergent (TE) immunization to RBC alloantigens through 28 ± 3 days after the last study transfusion.
Time Frame: From the start of the first study transfusion to 28 after the last study transfusion (between 29 and 35 days depending on the day of the last study transfusion).
Population: Participants who received at least one study transfusion with available data on the outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | INTERCEPT (Test) | Conventional (Control)
Number analyzed (Participants) | 159 | 162
Participants | 1 | 2

7. Other Pre Specified Outcome: Number of Participants With Transfusion Reactions (TR)
Description: Transfusion reactions (as defined by the CDC National Healthcare Safety Network) through 28 days after the last study transfusion
Time Frame: as for outcome 2
Population: Participants who received at least one study transfusion with available data on the outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | INTERCEPT (Test) | Conventional (Control)
Number analyzed (Participants) | 159 | 162
Participants | 4 | 0

8. Other Pre Specified Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Treatment-emergent SAEs through 28 days after the last study transfusion
Time Frame: as for outcome 2
Population: Participants who received at least one study transfusion with available data on the outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | INTERCEPT (Test) | Conventional (Control)
Number analyzed (Participants) | 159 | 162
Participants | 66 | 57

9. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Immunization to HLA Alloantigens Through 28 ± 3 Days From After the Last Study Transfusion
Description: Treatment emergent HLA Class 1 or Class 2 antibodies at high cutoff values
Time Frame: 28 days after the last study transfusion (between 29 and 35 days depending on the day of the last study transfusion).
Population: Data only available for a subset of subjects with samples collected both at baseline and Day 28, therefore only 114 INTERCEPT (Test) participants and 113 Conventional (Control) participants were available for analysis, as seen in Outcome Measure Data Table below.
Measure: Count of Participants; unit: Participants
Arm/Group | INTERCEPT (Test) | Conventional (Control)
Number analyzed (Participants) | 114 | 113
Participants
  HLA Class 1 | 17 | 13
  HLA Class 2 | 8 | 8

10. Other Pre Specified Outcome: Number of Participants With Treatment Emergent AEs Through 28 Days After the Last Study Transfusion.
Description: Treatment emergent adverse events through 28 days after the last study transfusion.
Time Frame: as for outcome 2
Population: Participants who received at least one study transfusion with available data on the outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | INTERCEPT (Test) | Conventional (Control)
Number analyzed (Participants) | 159 | 162
Participants | 153 | 147

ADVERSE EVENTS:
Time Frame: Adverse Events from the first study transfusion until 28 days following the last transfusion (29-35 days after the first transfusion). All cause mortality was assessed 75 days following the last transfusion (76-82 days after the first study transfusion).
Description: The number of participants at risk for adverse events includes all randomized subjects who received at least one study transfusion, based on the actual treatment received.
Arm/Group | INTERCEPT (Test) | Conventional (Control)
All-Cause Mortality (participants affected / at risk) | 13/159 | 10/162
Serious Adverse Events (participants affected / at risk) | 66/159 | 57/162
Other Adverse Events (participants affected / at risk) | 152/159 | 145/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INTERCEPT (Test) (N=159) | Conventional (Control) (N=162)
anaemia (Blood and lymphatic system disorders) | 2 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 4 | 2
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Arrhythmia (Cardiac disorders) | 1 | 1
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 8 | 2
Atrial flutter (Cardiac disorders) | 0 | 2
Atrioventricular block (Cardiac disorders) | 2 | 2
Atrioventricular block complete (Cardiac disorders) | 3 | 3
Bradyarrhythmia (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 4 | 4
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure acute (Cardiac disorders) | 2 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 3
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 2 | 4
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Coronary artery thrombosis (Cardiac disorders) | 1 | 0
Nodal rhythm (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 1
Pericardial haemorrhage (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Prosthetic cardiac valve thrombosis (Cardiac disorders) | 1 | 1
Right ventricular dysfunction (Cardiac disorders) | 1 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0
Sinus arrest (Cardiac disorders) | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular dysfunction (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 3 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal angiectasia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 4 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 2 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0
Effusion (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 2
Medical device site haemorrhage (General disorders) | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 7 | 2
Necrosis (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Hepatobiliary disorders (Hepatobiliary disorders) | 5 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 4 | 1
Liver injury (Hepatobiliary disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Corona virus infection (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 5
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 4
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Transfusion-related circulatory overload (Injury, poisoning and procedural complications) | 1 | 0
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 4 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 3 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 3 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 2
Nervous system disorder (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 15 | 3
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Renal infarct (Renal and urinary disorders) | 1 | 0
Renal injury (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Mediastinal haematoma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 | 12
Aortic thrombosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2
Haematoma (Vascular disorders) | 0 | 2
Haemorrhage (Vascular disorders) | 2 | 1
Hypoperfusion (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 6 | 2
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 1
Shock (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | INTERCEPT (Test) (N=159) | Conventional (Control) (N=162)
Anaemia (Blood and lymphatic system disorders) | 47 | 39
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 22 | 20
Leukocytosis (Blood and lymphatic system disorders) | 9 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 50 | 41
Atrial fibrillation (Cardiac disorders) | 35 | 54
Atrial flutter (Cardiac disorders) | 2 | 9
Nausea (Gastrointestinal disorders) | 9 | 8
Pyrexia (General disorders) | 6 | 11
Urinary tract infection (Infections and infestations) | 11 | 8
Procedural pain (Injury, poisoning and procedural complications) | 29 | 25
Transaminases increased (Investigations) | 6 | 9
Fluid overload (Metabolism and nutrition disorders) | 7 | 13
Hyperglycaemia (Metabolism and nutrition disorders) | 31 | 28
Hypocalcaemia (Metabolism and nutrition disorders) | 28 | 27
Hypokalaemia (Metabolism and nutrition disorders) | 22 | 24
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 | 12
Hypophosphataemia (Metabolism and nutrition disorders) | 21 | 23
Delirium (Psychiatric disorders) | 6 | 9
Acute kidney injury (Renal and urinary disorders) | 27 | 34
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 6 | 10
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 18 | 25
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 12
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 10
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 15 | 14
Hypertension (Vascular disorders) | 9 | 11
Hypotension (Vascular disorders) | 16 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT03459287/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT03459287/SAP_001.pdf
  • Informed Consent Form (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT03459287/ICF_002.pdf